CLINICAL TRIAL: NCT01222520
Title: An Eight-week Randomised Double-blind Study to Compare the Efficacy and Safety of Telmisartan 80 mg+ Amlodipine 5 mg Fixed-dose Combination vs. Telmisartan 80 mg Monotherapy in Patients With Hypertension Who Fail to Respond Adequately to Treatment With Telmisartan 80 mg Monotherapy
Brief Title: Telmisartan 80mg Non-responder Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1235.36
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Results first posted 2012-07-04 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — telmisartan amlodipine combination; Telmisartan

ARMS (2):
- Telmisartan and amlodipine FDC (Experimental): once a daily
  Interventions: Drug: Telmisartan and amlodipine
- Telmisartan monotherapy (Active Comparator): once a daily
  Interventions: Drug: Telmisartan

INTERVENTIONS:
Drug: Telmisartan and amlodipine — Telmisartan 80 mg and amlodipine 5 mg once a daily
  Arms: Telmisartan and amlodipine FDC
Drug: Telmisartan — 80 mg once a daily
  Arms: Telmisartan monotherapy

SUMMARY:
If a patient cannot have his or her blood pressure controlled with telmisartan 80 mg, an antihypertensive drug from different class should be started concomitantly.

In the Japanese 3x3 factorial trial of telmisartan and hydrochlorothiazide in essential hypertension patients whose diastolic blood pressure (DBP) are equal or more than 95 mmHg, the DBP control rate (less than 90 mmHg) after 8 weeks treatment of the telmisartan 80 mg monotherapy group (66 patients) was 41.5%. There should be medical needs of the telmisartan 80 mg and amlodipine 5 mg fixed dose combination because some patients cannot have his or her blood pressure controlled with telmisartan 80 mg.

Thus, this clinical trial is being conducted to evaluate the antihypertensive effect and safety of a fixed-dose combination (FDC) drug of 2 antihypertensive agents with different pharmacological effects, telmisartan 80 mg and amlodipine 5 mg (T80/A5 mg), compared with telmisartan 80 mg (T80 mg) monotherapy in Japanese patients with essential hypertension who fail to respond adequately to treatment with the maximum dose of telmisartan 80 mg monotherapy. In this trial, a multi-centre, randomised, double-blind, double-dummy, active-controlled, parallel group comparison method is employed.

ELIGIBILITY:
Inclusion criteria:

* Essential hypertensive patients

  * If already taking antihypertensive drugs, mean seated diastolic blood pressure (DBP) must be >=90 and >=114 mmHg
  * If not taking any antihypertensive drugs, mean seated DBP must be >=95 and >=114 mmHg
* Able to stop all current antihypertensive drugs without risk to the patient based on the investigators opinion.

Exclusion criteria:

* Patients taking 3 or more antihypertensive drugs at signing the informed consent form
* Patients with known or suspected secondary hypertension
* Patients with clinically relevant cardiac arrhythmia
* Congestive heart failure with New York Heart Association (NYHA) functional class III-IV
* Patients with recent cardiovascular events
* Patients with a history of stroke or transient ischaemic attack within last 6 months before signing the informed consent form
* Patients with a history of sudden deterioration of renal function with angiotensin II receptor blockers (ARBs) or angiotensin converting enzyme (ACE) inhibitors; or patients with post-renal transplant or post-nephrectomy
* Patients who have previously experienced characteristic symptoms of angioedema (such as facial, tongue, pharyngeal, or laryngeal swelling with dyspnea) during treatment with ARBs or ACE inhibitors
* Patients with known hypersensitivity to any component of the investigational product, or a known hypersensitivity to dihydropyridine-derived drugs
* Patients with hepatic and/or renal dysfunction
* Pre-menopausal women who are nursing or pregnant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (4):
- Japan (4):
  - 1235.36.01 Boehringer Ingelheim Investigational Site, Chuo-ku,Tokyo
  - 1235.36.04 Boehringer Ingelheim Investigational Site, Hiroshima, Hiroshima
  - 1235.36.02 Boehringer Ingelheim Investigational Site, Shinjuku-ku, Tokyo
  - 1235.36.03 Boehringer Ingelheim Investigational Site, Suita, Osaka

RESULTS

PARTICIPANT FLOW:
Period: Open-label run-in Period
Arm/Group | Telmisartan and Amlodipine FDC | Telmisartan
Started | 0 | 197
Completed | 0 | 174
Not Completed | 0 | 23
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Blood pressure criteria not met | 0 | 18
Not completed — Number of patients fulfilled | 0 | 3
Period: Double-blind Period
Arm/Group | Telmisartan and Amlodipine FDC | Telmisartan
Started | 87 | 87
Completed | 86 | 85
Not Completed | 1 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Study medication stolen | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telmisartan and Amlodipine FDC | Telmisartan | Total
Number analyzed (Participants) | 87 | 87 | 174
Age, Continuous [Mean (Standard Deviation); unit: year] | 54.5 (9.0) | 54.8 (8.6) | 54.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 13 | 33
  Male | 67 | 74 | 141

OUTCOME MEASURES:

1. Primary Outcome: Reduction From the Reference Baseline in Mean Seated Diastolic Blood Pressure (DBP) at Trough
Description: Reference baseline: Status of patients after the 8-week open-label run-in period with telmisartan monotherapy, where patients' eligibility to enter the double-blind treatment period was examined At trough: 24-hour post-dosing
Time Frame: Baseline, 8 weeks
Population: Full analysis set (FAS)
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan and Amlodipine FDC | Telmisartan
Number analyzed (Participants) | 87 | 86
mmHg | 12.28 (0.73) | 3.14 (0.74)
Statistical Analysis 1: Comparison: Telmisartan and Amlodipine FDC vs Telmisartan; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least square mean difference = 9.14, 95% CI [7.09 to 11.18]

2. Secondary Outcome: Reduction From the Reference Baseline in Mean Seated Systolic Blood Pressure (SBP) at Trough
Description: as for outcome 1
Time Frame: Baseline, 8 weeks
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan and Amlodipine FDC | Telmisartan
Number analyzed (Participants) | 87 | 86
mmHg | 18.37 (1.10) | 3.49 (1.10)
Statistical Analysis 1: Comparison: Telmisartan and Amlodipine FDC vs Telmisartan; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least square mean difference = 14.88, 95% CI [11.82 to 17.94]

3. Secondary Outcome: Seated DBP Control Rate at Trough
Description: DBP control rate: The rate of patients with controlled seated DBP at trough of less than 90 mmHg after the 8-week double-blind period At trough: 24-hour post-dosing
Time Frame: 8 weeks
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Telmisartan and Amlodipine FDC | Telmisartan
Number analyzed (Participants) | 87 | 86
Percentage of participants
  No | 29.9 | 73.3
  Yes | 70.1 | 26.7
Statistical Analysis 1: Comparison: Telmisartan and Amlodipine FDC vs Telmisartan; Test type: Superiority or Other; p < 0.0001, Fisher Exact

4. Secondary Outcome: Seated SBP Control Rate at Trough
Description: SBP control rate: The rate of patients with controlled seated SBP at trough of less than 140 mmHg after the 8-week double-blind period At trough: 24-hour post-dosing
Time Frame: 8 weeks
Population: Patients included in FAS and with seated SBP ≥140 mmHg at reference baseline
Measure: Number; unit: Percentage of participants
Arm/Group | Telmisartan and Amlodipine FDC | Telmisartan
Number analyzed (Participants) | 50 | 52
Percentage of participants
  No | 26.0 | 71.2
  Yes | 74.0 | 28.8
Statistical Analysis 1: Comparison: Telmisartan and Amlodipine FDC vs Telmisartan; Test type: Superiority or Other; p < 0.0001, Fisher Exact

5. Secondary Outcome: Seated DBP Response Rate at Trough
Description: DBP response rate: The rate of patients who achieved an adequate response in seated DBP at trough (<90 mmHg and/or reduction from reference baseline ≥10 mmHg) after the 8-week double-blind period At trough: 24-hour post-dosing
Time Frame: 8 weeks
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Telmisartan and Amlodipine FDC | Telmisartan
Number analyzed (Participants) | 87 | 86
Percentage of participants
  No | 19.5 | 69.8
  Yes | 80.5 | 30.2
Statistical Analysis 1: Comparison: Telmisartan and Amlodipine FDC vs Telmisartan; Test type: Superiority or Other; p < 0.0001, Fisher Exact

6. Secondary Outcome: Seated SBP Response Rate at Trough
Description: SBP response rate: The rate of patients who achieved an adequate response in seated SBP at trough (<140 mmHg and/or reduction from reference baseline ≥20 mmHg) after the 8-week double-blind period At trough: 24-hour post-dosing
Time Frame: 8 weeks
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Telmisartan and Amlodipine FDC | Telmisartan
Number analyzed (Participants) | 87 | 86
Percentage of participants
  No | 11.5 | 48.8
  Yes | 88.5 | 51.2
Statistical Analysis 1: Comparison: Telmisartan and Amlodipine FDC vs Telmisartan; Test type: Superiority or Other; p < 0.0001, Fisher Exact

7. Secondary Outcome: Seated Blood Pressure (BP) Normalisation at Trough
Description: Seated blood pressure (BP) normalisation: The numbers of patients whose blood pressure was within normalisation criterion in terms of seated blood pressure after the 8-week double-blind period At trough: 24-hour post-dosing
Time Frame: 8 weeks
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Telmisartan and Amlodipine FDC | Telmisartan
Number analyzed (Participants) | 87 | 86
Participants
  No | 28 | 66
  Optimal | 21 | 2
  Normal | 22 | 7
  High-normal | 16 | 11
Statistical Analysis 1: Comparison: Telmisartan and Amlodipine FDC vs Telmisartan; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: From drug administration in the double blind treatment period until 24 hours after the last dosing, up to 63 days.
Arm/Group | Telmisartan and Amlodipine FDC | Telmisartan
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/87
Other Adverse Events (participants affected / at risk) | 5/87 | 2/87
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telmisartan and Amlodipine FDC (N=87) | Telmisartan (N=87)
Nasopharyngitis (Infections and infestations) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.